CLINICAL TRIAL: NCT04756492
Title: Prognostic Factors for Treatment Responses in Patients With Active Lupus Nephritis at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Helmy, assistant lecture, Sohag University
Other Study IDs: Soh-Med-21-02-06
Record Dates: First submitted 2021-02-14; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: We Aim to Examine the Predictors of Sustained Complete Renal Remission in Patients With Lupus Nephritis at Sohag University Hospital
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: sandimmun — follow up for treatment response
  Other Names: indoxan

SUMMARY:
Systemic lupus erythematosus (SLE) is an autoimmune disease which may give rise to multiple organ involvement because of immune complex deposits. Lupus nephritis (LN) is one of the severe manifestations of systemic lupus erythematous (SLE) and a common cause for end-stage renal disease, significantly affecting the survival of SLE patients Immunosuppressive treatment is the major therapy for active LN. Generally, at least six months are needed to assess treatment responses Failure to respond to immunosuppressive therapy can lead to a worsening of renal function

DETAILED DESCRIPTION:
This study will be prospectively analyzing the clinical data of LN patients who received standard immunosuppressive therapy and were regularly followed up at our center for more than six months. These patients will not change treatment regimen during the six months.

As remission is an independent predictor of good long term prognosis in lupus nephritis. We aim to examine the predictors of sustained complete renal remission in patients with lupus nephritis at Sohag University Hospital and to analyze data of lupus nephritis patients to find parameters that can predict remission and improve outcome of our cases

ELIGIBILITY:
Inclusion Criteria:

* o Patients diagnosed with LN at Sohag University Hospital

  * Patients in regular follow-up for more than six months after immunosuppressive therapy
  * Baseline urinary protein/creatinine ratio (UPCR) more than 1 g/g
  * Baseline C3 less than 55 mg/ dl
  * No change in immunosuppressive therapy within six months

Exclusion Criteria:

* o Patients with incomplete pathological data and the number of glomeruli being <10 per biopsy specimen

  * Age <14 years old End-stage renal disease (ESRD) status on admission (sustained estimated glomerular filtration rate (eGFR) <15 ml/min per 1.73m2)
  * Patients with advanced comorbid conditions like advanced liver cirrhosis or heart failure or malignancy

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: o Patients diagnosed with LN at Sohag University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
complete renal response | 6 months
  Alb _35 g/l, UPCR<0.3 g/g, a normal range of sCr or at a level increasing no more than 15% from baseline and without lupus flares.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
sharing final results only